CLINICAL TRIAL: NCT02432976
Title: Impact of Intravenous Exenatide Versus Insulin on Quality of Life in Cardiac Surgery Patients: an Ancillary Study of the ExSTRESS Phase II/III Clinical Trial
Brief Title: Impact of Perioperative Exenatide Infusion on Quality of Life in Cardiac Surgery Patients
Acronym: ExeQOL
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Collaborators: AstraZeneca (Industry); Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09/503
Record Dates: First submitted 2015-04-29; First posted 2015-05-04 (Estimated); Last update posted 2021-03-09 (Actual); Status verified 2016-01

CONDITIONS: Quality of Life
Keywords: Quality of Life; Cardiac Surgery; Coronary Artery Bypass Graft Surgery; Incretin mimetic; Exenatide
MeSH Terms: interventions — Exenatide; Incretins; Insulin; Insulin Lispro; purine-analog-sensitive kinase, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exenatide group (Experimental): Exenatide. Exenatide: bolus of 0.05 µg/min infused during the 1st hour of treatment, followed by a continuous infusion of 0.025 µg/min until the end of treatment.
  The exenatide therapy will begin as soon as a blood glucose level is above 140 mg/dl will be measured. A of exenatide will be intravenously .
  The treatment will be administrated during the first postoperative 48 hours in the intensive care unit or until intensive care unit discharge if this event occurs earlier.
  Interventions: Drug: Exenatide
- Insulin group (Active Comparator): Insulin: Humalog (insulin lispro human analog). The insulin therapy will begin as soon as a blood glucose level is above 140 mg/dl will be measured.
  The dose of insulin intravenously infused will be adapted to blood glucose measurements, following the insulin therapy protocol used in our department.
  The insulin therapy protocol used in our department and prescribed as the benchmark treatment in the present study has been validated in a previous study. It has been derived from the protocol validated by Goldberg et al.
  Interventions: Drug: Insulin

INTERVENTIONS:
Drug: Exenatide — Exenatide. Exenatide: bolus of 0.05 µg/min infused during the 1st hour of treatment, followed by a continuous infusion of 0.025 µg/min until the end of treatment.
  The exenatide therapy will begin as soon as a blood glucose level is above 140 mg/dl will be measured. A of exenatide will be intravenously .
  The treatment will be administrated during the first postoperative 48 hours in the intensive care unit or until intensive care unit discharge if this event occurs earlier.
  Other Names: Byetta; Exendin-4; Incretin
  Arms: Exenatide group
Drug: Insulin — Insulin: Humalog (insulin lispro human analog). The insulin therapy will begin as soon as a blood glucose level is above 140 mg/dl will be measured.
  The dose of insulin intravenously infused will be adapted to blood glucose measurements, following the insulin therapy protocol used in our department.
  The insulin therapy protocol used in our department and prescribed as the benchmark treatment in the present study has been validated in a previous study. It has been derived from the protocol validated by Goldberg et al.
  Other Names: Humalog; Insulin Lispro; Human Analog
  Arms: Insulin group

SUMMARY:
A diminution of quality of life is often reported by patients after coronary artery bypass graft (CABG) surgery. A part of this diminution could be explain by postoperative left ventricular (LV) dysfunction.

Exenatide (Byetta®) is an incretin mimetic, characterized by an anti-hyperglycemic effect that depends on the blood glucose level. Recent data have suggested that exenatide could improve LV function by an inotropic effect in patients suffering from cardiogenic shock or from congestive heart failure. Moreover, patients suffering from congestive heart failure reported a better quality of life when they were treated with exenatide compared to placebo.

The investigators hypothesize that perioperative exenatide infusion could improve postoperative quality of life in CABG surgery patients.

DETAILED DESCRIPTION:
The ExeQOL study is an ancillary study of the ExSTRESS trial (www.clinicaltrials.gov identifier: NCT01969149).

The ExSTRESS trial is a phase II/III randomized-controlled trial that aim at assessing intravenous exenatide versus insulin for perioperative glycemic control in CABG surgery.

The phase II of the ExStress trial will assess the safety and the efficacy of a continuous intravenous infusion of exenatide for the management of post operative stress hyperglycemia after planned coronary artery graft bypass (CABG) surgery.

The aim of the phase III of the ExSTRESS trial is to compare the efficacy of a continuous intravenous infusion of exenatide to the gold standard treatment, i.e the intravenous infusion of short-acting insulin, for the management of post operative stress hyperglycemia after planned CABG surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18.
* Patient consent.
* Non insulin requiring type 2 diabetic patients.
* Non diabetic patients.
* Planned coronary artery bypass graft (CABG) surgery.
* ASA (American Society of Anesthesiologists) score 1, 2, or 3.

Exclusion Criteria:

* Pregnancy and breast feeding.
* Pancreatectomy.
* Acute pancreatitis.
* Chronic pancreatitis.
* Type 1 diabetic patients.
* Insulin requiring type 2 patients.
* HbA1c>8%
* Ketoacidosis.
* Hyperosmolar coma.
* Preoperative blood glucose level above 300 mg/dl [21].
* Insulin or exenatide contraindication.
* History of renal transplantation or currently receiving renal dialysis or creatinine clearance below 60 ml/min.
* Emergency surgery.
* Planned non CABG cardiac surgery.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2015-05; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Variation of the SF-36 score value at 3-months | 3 months
  The SF-36 score is a self-administered questionnaire that assess both the physical and the psychosocial health-related quality of life.
  The use of the SF-36 score is recommended by the French Health Authority in coronary patients.
  The variation of the SF-36 score value at 3-months is defined as the difference between the SF36-score value at 3 months minus the preoperative SF-36 score value.

SECONDARY OUTCOMES:
Variation of the SF-36 score value at 1-month | 1 month
  The SF-36 score is a self-administered questionnaire that assess both the physical and the psychosocial health-related quality of life.
  The use of the SF-36 score is recommended by the French Health Authority in coronary patients.
  The variation of the SF-36 score value at 1-month is defined as the difference between the SF36-score value at 1 month minus the preoperative SF-36 score value.
Variation of the SF-36 score value at 6-months | 6 months
  The SF-36 score is a self-administered questionnaire that assess both the physical and the psychosocial health-related quality of life.
  The use of the SF-36 score is recommended by the French Health Authority in coronary patients.
  The variation of the SF-36 score value at 6-months is defined as the difference between the SF36-score value at 6 months minus the preoperative SF-36 score value.
Variation of the SF-36 score value at 12-months | 12 months
  The SF-36 score is a self-administered questionnaire that assess both the physical and the psychosocial health-related quality of life.
  The use of the SF-36 score is recommended by the French Health Authority in coronary patients.
  The variation of the SF-36 score value at 12-months is defined as the difference between the SF36-score value at 12 months minus the preoperative SF-36 score value.
1-month mortality | 1 month
3-months mortality | 3 months
6-months mortality | 6 month
12-months mortality | 12 months
Postoperative left ventricular function | Day 7
  Left ventricular function will be assessed during a transthoracic echocardiography performed at Day 7.
  Left ventricular ejection fraction and filling pressure will be measured during this procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume BESCH, M.D., Principal Investigator — CHRU Besançon; Sebastien PILI-FLOURY, M.D., PhD, Study Director — CHRU Besançon
Locations (1):
- Post operative intensive care unit of the cardiac surgery department, Besançon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Goldberg PA, Sakharova OV, Barrett PW, Falko LN, Roussel MG, Bak L, Blake-Holmes D, Marieb NJ, Inzucchi SE. Improving glycemic control in the cardiothoracic intensive care unit: clinical experience in two hospital settings. J Cardiothorac Vasc Anesth. 2004 Dec;18(6):690-7. doi: 10.1053/j.jvca.2004.08.003. PMID 15650975
- [Background] Studer C, Sankou W, Penfornis A, Pili-Floury S, Puyraveau M, Cordier A, Etievent JP, Samain E. Efficacy and safety of an insulin infusion protocol during and after cardiac surgery. Diabetes Metab. 2010 Feb;36(1):71-8. doi: 10.1016/j.diabet.2009.05.008. Epub 2010 Jan 25. PMID 20097589
- [Background] Perneger TV, Leplege A, Etter JF, Rougemont A. Validation of a French-language version of the MOS 36-Item Short Form Health Survey (SF-36) in young healthy adults. J Clin Epidemiol. 1995 Aug;48(8):1051-60. doi: 10.1016/0895-4356(94)00227-h. PMID 7775992
- [Background] Sokos GG, Nikolaidis LA, Mankad S, Elahi D, Shannon RP. Glucagon-like peptide-1 infusion improves left ventricular ejection fraction and functional status in patients with chronic heart failure. J Card Fail. 2006 Dec;12(9):694-9. doi: 10.1016/j.cardfail.2006.08.211. PMID 17174230
- [Background] Sokos GG, Bolukoglu H, German J, Hentosz T, Magovern GJ Jr, Maher TD, Dean DA, Bailey SH, Marrone G, Benckart DH, Elahi D, Shannon RP. Effect of glucagon-like peptide-1 (GLP-1) on glycemic control and left ventricular function in patients undergoing coronary artery bypass grafting. Am J Cardiol. 2007 Sep 1;100(5):824-9. doi: 10.1016/j.amjcard.2007.05.022. Epub 2007 Jun 14. PMID 17719327
- See also: Link to ExStress Study protocol — https://clinicaltrials.gov/ct2/show/NCT01969149?term=exstress&rank=1